CLINICAL TRIAL: NCT06555276
Title: Post-market Clinical Follow-up of Disposable Endoscope Linear Cutting Staplers and Components
Status: Not yet recruiting | Type: Observational
Sponsor: Suzhou Kerui Medical Technology Co., Ltd (Other)
Collaborators: Jiangsu Channel Medical Device Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: CN-ED-CTP
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Gastric Disease
Keywords: stapler; anastomosis
MeSH Terms: conditions — Stomach Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Disposable endoscope linear cutting stapler and components — to use the study device for excision, transection and anastomosis of lung, bronchial tissue, stomach and intestine in open or endoscopic surgery.

SUMMARY:
This is a multi-center and retrospective cohort study to evaluate the efficacy and safety of disposable linear cutting staplers and components in soft tissue resection, transection and anastomosis.

DETAILED DESCRIPTION:
The disposable endoscopic linear cutting staplers and components developed and produced by Jiangsu Channel Medical Device Co., Ltd. can be used in open or endoscopic surgery of lung, bronchial tissue, stomach and intestine resection, transection and anastomosis. They have been registered in China for many years and have been widely used, and have been certified by the European Union in 2021. The number is CIM.2021.106.14629. This study intends to conduct a multi-center retrospective cohort study in China, collect clinical application data of Chinese patients, conduct statistical analysis on the clinical application data, confirm whether the expected effectiveness and safety are achieved, and further extrapolate to the EU population.

ELIGIBILITY:
Inclusion Criteria:

* gender unlimited, age unlimited ② open or endoscopic surgery ③ resection, transection and anastomosis of lung, bronchial tissue, stomach and intestines.

  * use the study device during surgery

Exclusion Criteria:

* patients with contraindications to the product, such as severe mucosal edema, operation of the hemostatic site that cannot be observed, or off-label use of the liver and spleen;

  * combined with other similar products (staplers) for surgical site excision, transsection and anastomosis; ③ surgical records are incomplete, and information related to major indicators cannot be extracted; ④ other situations that the researcher considers inappropriate for inclusion in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who need open or endoscopic surgery using the study device for resection, transection and anastomosis for liver, bronchial tissue, stomach and intestines. Those who meet the inclusion criteria and don't meet the exclusion criteria will be enrolled.
Sampling Method: Probability Sample
Enrollment: 195 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
anastomosis success rate | within six months after surgery
  According to surgical records and hospitalization records, the condition of no reoperation in situ was defined as successful anastomosis. Anastomosis success rate=cases of successful anastomosis/total cases of surgery ×100%

CONTACTS AND LOCATIONS:
Overall Officials: zhengliang Tu, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No